CLINICAL TRIAL: NCT04482569
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled Sequential Group Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of XNW4107 for Injection, and Multiple Doses of XNW4107 for Injection in Combination With Imipenem/Cilastatin for Injection in Healthy Adult Male Subjects
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics of XNW4107 Alone or in Combination With Imipenem/Cilastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: XNW4107-001
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Infections
Keywords: XNW4107; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose Study (Experimental): Six XNW4107 doses ( 50-1250 mg ), each administered as a single dose with 60-minute IV infusion
  Interventions: Drug: XNW4107
- Multiple Ascending Dose Study (Experimental): Three XNW4107 doses (167-500 mg), each administered as 60-minute IV infusion every 6 hours for 7 days
  Interventions: Drug: XNW4107
- Multiple Dose Study of XNW4107 +Imipenem/Cilastatin (Experimental): 500 mg XNW4107 co-administered with imipenem/cilastatin as 60-minute IV infusion every 6 hours for 14 days
  Interventions: Drug: XNW4107

INTERVENTIONS:
Drug: XNW4107 — Single or multiple dose ascending study for XNW4107 alone or multiple dose study of XNW4107 in combination with imipenem/cilastatin

SUMMARY:
This is a 3-part, first-in-human study to evaluate the safety, tolerability and pharmacokinetics of escalating doses of XNW4107 given as intravenous (IV) infusion in healthy male subjects. In part 1, subjects will receive a single dose of XNW4107. In part 2, subjects will receive XNW4107 for 7 days. In Part 3, subjects will receive XNW4107 in combination with imipenem/cilastatin for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged 18-65 years
* Body Mass Index (BMI) between 18.5 - 32.0, inclusive.
* In good general health, as determined by the Investigator, based on medical history, physical examination, 12 lead electrocardiogram (ECG), vital sign (VS) measurements, and laboratory test results.
* Normal blood pressure (BP), defined as: systolic BP (SBP) ≥90 mmHg and ≤140 mmHg; and diastolic BP (DBP) <90 mmHg at the time of Screening
* Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subject) in addition to an acceptable method (female partner) of contraception for the duration of the study and for at least 90 days post last dose.
* Negative serology results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus antibody (HIV Ab), hepatitis E immunoglobulin M antibody (IgM anti HEV), and Treponema pallidum antibody chemiluminescent immunoassay (TP IA).
* Negative serology results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus antibody (HIV Ab), hepatitis E immunoglobulin M antibody (IgM anti HEV), and Treponema pallidum antibody chemiluminescent immunoassay (TP IA).
* Non smoker (with no use of other tobacco or nicotine containing products, in any form), as documented by history (no nicotine within 3 months prior to Screening)
* Negative results for drugs of abuse, alcohol, and cotinine at Screening and Admission

Exclusion Criteria:

* History of clinically significant psychiatric disorder within the past 5 years.
* History of stroke, chronic seizures, or other major neurological disorder.
* History or evidence of drug/alcohol abuse within 1 year prior to Screening.
* History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or disease.
* History of cancer (malignancy).
* History of any illness that, in the opinion of the study investigator, may confound the results of the study or pose additional risk to the subject if he participates in the study.
* Administration of another investigational medication within 30 days (or 5 half lives, whichever is longer) prior to study drug administration.
* Participation in an investigational device study within 30 days prior to study drug administration.
* Excessive consumption of alcohol, defined as >3 alcoholic beverages per day (10 ounces of beer [284 mL], 4 ounces of wine [125 mL], or 1 ounce of distilled spirits [25 mL] is approximately equivalent to 1 alcoholic beverage)
* Excessive consumption of coffee, tea, cola, or other caffeinated beverages; excessive consumption is defined as >6 servings per day (1 serving contains approximately 120 mg caffeine)
* History and/or family history of congenital long QT syndrome, unexplained syncope, or other additional risks of Torsade de Pointes or sudden premature death.
* Any ECG abnormality considered to be clinically significant by the principal investigator (PI)/designee;
* Glomerular filtration rate (GFR) ≤80 mL/min/1.73 m2, as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation.
* Ongoing liver disease or unexplained liver function test (LFT) elevations
* History of hypersensitivity to β lactam antibiotics (including, but not limited to imipenem)
* History of significant multiple and/or severe allergies (including latex allergy);
* Loss or donation of blood (approximately 500 mL) within 60 days prior to study drug administration on Day 1, or donation of bone marrow or peripheral stem cells within 90 days prior to study drug administration on Day 1.
* History of infectious disease within 28 days prior to study drug administration on Day 1 that, in the opinion of the investigator, would affect the subject's ability to participate in the trial.
* Venous access considered inadequate for PK sample collection and IV infusion; history or evidence of adverse symptoms associated with IV access, phlebotomy, or blood donation.
* Employee or family member of the investigator, study site personnel, or sponsor.
* Any other clinically relevant abnormality in the opinion of the investigators from the following: medical and/or surgical history, physical examination, vital signs, 12-lead ECG, serum chemistry, hematology, and urinalysis.
* Any other reason that, in the opinion of the investigator, would render the subject unsuitable for study enrollment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by number of participants experiencing adverse events | Change from baseline up to day 43 post-intervention
  Number of participants who experience adverse events in different grades, as defined by Common Terminology for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jason Le, Study Chair — Evopoint Biosciences Inc.
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States